CLINICAL TRIAL: NCT04695743
Title: Virtual CST - A Collaborative Proof of Concept Study With FaceCog HK in Response to the Covid-19 Pandemic
Brief Title: Group CST Using Zoom: A Proof of Concept Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17127/002
Record Dates: First submitted 2020-12-11; First posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2021-01

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Attendance at online CST groups
  Interventions: Other: Online Cognitive Stimulation Therapy
- Control (No Intervention): Treatment as usual

INTERVENTIONS:
Other: Online Cognitive Stimulation Therapy — Participants will attend 14 x 1 hour online CST sessions that involve a variety of activities to stimulate the brain and focus on cognitive strengths based on a variety of themes i.e. childhood, using money, etc. This will aim to be multisensory and give choice and empowerment to participants. Benefits of face to face CST are shown to slow cognitive decline and improve quality of life. Adapting it for online use will investigate whether participants can still benefit in this way.
  Arms: Intervention

SUMMARY:
People living with dementia (PLWD) often struggle to access services and treatment which may benefit their emotional and cognitive wellbeing, as well as disease progression. Transport provision; hospital access and restricted mobility are barriers that often deny people the opportunity to receive treatment in-line with NICE guidelines. Considering the current Covid-19 pandemic, hospital access and face-to-face treatment is even more limited at present; with services across the UK unable to offer their usual levels of care and support. This is particularly the case for people in vulnerable groups. Therefore, many services have been considering the potential of remote-access therapy, specifically the use of video-conferencing apps. During the covid-19 crisis and beyond, it is of urgent and practical need that we develop more accessible, innovative home-based group interventions to people with dementia that can be delivered remotely. A group at The University of Hong Kong, are undertaking a study entitled 'FaceCog' which involves the delivery of Cognitive Stimulation Therapy (CST) via the video-conferencing application 'Zoom'. CST is an established, evidence-based group intervention shown to improve quality of life and slow down cognitive deterioration in PLWD. In collaboration with the Hong Kong 'FaceCog' team, we propose to deliver a culturally adapted version of their Zoom-CST protocol in the UK in a proof of concept study during the current Covid-19 pandemic. The facecog Zoom-CST protocol is the first virtual CST protocol of its kind that we are aware of. It closely follows the original, evidence-based CST manual that was developed in the UK. It has been slightly adapted to make it useable on a virtual platform and to be culturally sensitive for use in Hong Kong. It incorporates all key elements and principles that have been evidenced to make the treatment effective. As we are delivering it in the UK, we will be using activities from the original manual, in place of the activities that have been adapted for the Hong Kong protocol. For example, we will use British phrases in the word games session rather than Chinese proverbs.

Data on recruitment, attrition, attendance data, focus groups, participant-completed session feedback forms and qualitative post-session interviews, will offer us the opportunity to assess intervention acceptability. Outcomes related to cognition, quality of life and mood will allow us to make inferences about the potential for clinical impacts of such an intervention. Engagement analysis will allow us to explore the potential barriers and facilitators to virtual-delivered CST for this population and highlight any potential adaptations to intervention which may be needed. This project is intended as a preliminary exploration which will pave the way for future intervention-modifications and pilot-studies which can evaluate the potential benefits of 'virtually'-delivered CST.

This research aims to:

* Modify a pre-existing Zoom-CST protocol (FaceCog HK) to be culturally relevant and deliverable remotely within the UK.
* Modify and develop resources for the groups, along with dementia-friendly 'how to' guides on using the chosen video-conferencing application.
* Consult with stakeholders (including staff working within dementia care - clinical staff, charity organisations, and PLWD and their carers) about the potential foreseen barriers and facilitators to successful implementation of virtual-CST. Two remote, 'virtual' focus groups are proposed, one for professionals, and one for PLWD and/or informal carers.
* Asses virtual CST's feasibility as guided by Orsmond and Cohn's (2015) discussion article on this topic, which identifies objectives of feasibility studies as, an evaluation of recruitment capability and sample characteristics, data collection procedures and outcome measures, the acceptability and suitability of the intervention and study procedures, the resources and ability to manage and implement the study and intervention, participants' responses to the intervention.

ELIGIBILITY:
Inclusion criteria:

* Must have a clinical diagnosis of dementia and be within the 'mild-moderate' stages of disease progression.
* Must be able to communicate verbally in English.
* Must have capacity to consent to complete measures and to consent to video recording of the individual sessions.
* Must have access to a device capable of video-conferencing and internet at home.
* Must not be accessing any other psychosocial intervention (I.e. psychological therapy) at the time of participation

Exclusion criteria

* Not having a clinical diagnosis of dementia or being within the 'moderate- sever' stages of disease progression
* Not being able to communicate verbally in English
* Not have the capacity to take consent to participation
* Not have access to a device capable of video-conferencing and internet at home.
* If the person is accessing any other psychosocial intervention (I.e. psychological therapy) at the time of participation

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
ADAS-Cog (adapted for virtual use) - change is being assessed | To be completed within one week before and within one week after the intervention
  Assessment of cognitive skills, used in dementia research
MOCA blind- change is being assessed | To be completed within one week before and within one week after the intervention
  Cognitive screening tool
Geriatric Depression Scale- change is being assessed | To be completed within one week before and within one week after the intervention
  Screen for depression in older adults
QoL-AD- change is being assessed | To be completed within one week before and within one week after the intervention
  Quality of Life questionnaire for use in dementia

SECONDARY OUTCOMES:
Post intervention interviews | Within 1 month post intervention
  Qualitative date on experiences from the group

CONTACTS AND LOCATIONS:
Locations (1):
- University College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No